CLINICAL TRIAL: NCT03168815
Title: Low-Flow vs. High-Flow Nasal Cannula for Hypoxemic Immunocompromised Patients During Diagnostic Bronchoscopy: A Randomized Controlled Trial
Brief Title: Low-Flow vs. High-Flow Nasal Cannula for Hypoxemic Immunocompromised Patients During Diagnostic Bronchoscopy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Principal Investigator, Sangeeta Mehta, Professor, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: vSep2016
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Immunocompromised; Hematologic Malignancy; Post Hematopoietic Stem Cell Transplant; Hypoxia; Pulmonary Infiltrates
Keywords: HFNC; Bronchoscopy; Hypoxia; Immunocompromised; Hematological malignancy
MeSH Terms: conditions — Hematologic Neoplasms; Hypoxia

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either HFNC delivered at 50 L/min with FiO2 50% delivered for at least 5 min prior to FOB and throughout the procedure; or to conventional supplemental LFNC delivered at 6L/min applied for at least 5 minutes prior to FOB and throughout the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Flow Nasal Cannula (HFNC) (Experimental): Oxygen is delivered at 50 L/min with FiO2 50% delivered for at least 5 min prior to FOB and throughout the procedure.
  Interventions: Device: High Flow Nasal Cannula or Low Flow Nasal Cannula
- Low Flow Nasal Cannula (LFNC) (Active Comparator): Oxygen is delivered at 6L/min applied for at least 5 minutes prior to FOB and throughout the procedure.
  Interventions: Device: High Flow Nasal Cannula or Low Flow Nasal Cannula

INTERVENTIONS:
Device: High Flow Nasal Cannula or Low Flow Nasal Cannula — HFNC vs LFNC

SUMMARY:
Pneumonia is a lung infection. Fiberoptic bronchoscopy is a test to diagnose the type of lung infection. While this procedure is being performed, a small amount of oxygen is delivered into the nose (low flow nasal cannula). Occasionally during this procedure, the blood oxygen of the patient may drop and an intervention such as increasing the oxygen flow, or placing the patient on a breathing machine is required. An alternative device called 'Optiflow' can provide high flow oxygen through nasal cannula, and is comfortable for patients. If Optiflow is used during bronchoscopy, it may prevent the blood oxygen from dropping.

DETAILED DESCRIPTION:
Pneumonia is a lung infection that is a common complication in people with cancer, because of a weak immune system. Fiberoptic bronchoscopy is a test that is commonly used to help doctors diagnose the type of lung infection and treat it appropriately. It involves passing a thin tube with a camera at the end inside the lungs, and taking some fluid samples which are sent for analysis. While this procedure is being performed, a small amount of oxygen is delivered into the nose (low flow nasal cannula). Occasionally during this procedure, the blood oxygen of the patient may drop (even if the patient is receiving oxygen, and especially if the patient has severe pneumonia), and the procedure may have to be interrupted or prematurely stopped. If the oxygen level drops significantly, an intervention such as increasing the oxygen flow, or in the worst-case scenario temporarily placing the patient on a breathing machine is required. An alternative device called 'Optiflow' can provide high flow oxygen through nasal cannula, and is comfortable for patients. Optiflow was approved by Health Canada in 2006, and is commonly used in hospitals in Ontario and around the world to support patients whose blood oxygen is low. If Optiflow is used during bronchoscopy, it may prevent the blood oxygen from dropping.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years scheduled to undergo FOB (as determined by their medical care team) who are immunocompromised (active hematologic malignancy or post hematopoietic stem cell transplant), and are hypoxic with pulmonary infiltrates. Hypoxia will be defined as requiring supplemental low flow oxygen ≥ 2L/min by nasal cannula to maintain SpO2 >90%.

Exclusion Criteria:

1. requiring supplemental oxygen > 8L/min by nasal cannula;
2. receiving HFNC before randomization;
3. nasal deformity or packing precluding HFNC use;
4. hypercapnia (PaCO2 > 60) or respiratory acidosis (pH <7.25);
5. requiring NIV for over 1 hour or intubated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Desaturation during FOB | The SpO2 will be measured using a bedside SpO2 measuring device during or 1 hour post-FOB defined as a drop in SpO2 of 4% or more for > 1 minute or any drop in O2 <90% necessitating an increase in FiO2 to maintain a saturation ≥92% for at least 1 minute.
  Any desaturation during FOB or during the 1 hour post-FOB defined as a drop in SpO2 of 4% or more for more than 1 minute or any drop in O2 less than 90%, and necessitating an increase in FiO2 to maintain a saturation ≥92% for at least 1 minute.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sangeeta Mehta, MD, FRCPC, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hummel M, Rudert S, Hof H, Hehlmann R, Buchheidt D. Diagnostic yield of bronchoscopy with bronchoalveolar lavage in febrile patients with hematologic malignancies and pulmonary infiltrates. Ann Hematol. 2008 Apr;87(4):291-7. doi: 10.1007/s00277-007-0391-6. Epub 2007 Oct 12. PMID 17932672
- [Background] Shannon VR, Andersson BS, Lei X, Champlin RE, Kontoyiannis DP. Utility of early versus late fiberoptic bronchoscopy in the evaluation of new pulmonary infiltrates following hematopoietic stem cell transplantation. Bone Marrow Transplant. 2010 Apr;45(4):647-55. doi: 10.1038/bmt.2009.203. Epub 2009 Aug 17. PMID 19684637
- [Background] Kuehnhardt D, Hannemann M, Schmidt B, Heider U, Possinger K, Eucker J. Therapeutic implication of BAL in patients with neutropenia. Ann Hematol. 2009 Dec;88(12):1249-56. doi: 10.1007/s00277-009-0747-1. Epub 2009 May 5. PMID 19415277
- [Background] Hohenadel IA, Kiworr M, Genitsariotis R, Zeidler D, Lorenz J. Role of bronchoalveolar lavage in immunocompromised patients with pneumonia treated with a broad spectrum antibiotic and antifungal regimen. Thorax. 2001 Feb;56(2):115-20. doi: 10.1136/thorax.56.2.115. PMID 11209099
- [Background] Goldstein RA, Rohatgi PK, Bergofsky EH, Block ER, Daniele RP, Dantzker DR, Davis GS, Hunninghake GW, King TE Jr, Metzger WJ, et al. Clinical role of bronchoalveolar lavage in adults with pulmonary disease. Am Rev Respir Dis. 1990 Aug;142(2):481-6. doi: 10.1164/ajrccm/142.2.481. PMID 2200319
- [Background] Matsushima Y, Jones RL, King EG, Moysa G, Alton JD. Alterations in pulmonary mechanics and gas exchange during routine fiberoptic bronchoscopy. Chest. 1984 Aug;86(2):184-8. doi: 10.1378/chest.86.2.184. PMID 6744959
- [Background] Schnabel RM, van der Velden K, Osinski A, Rohde G, Roekaerts PM, Bergmans DC. Clinical course and complications following diagnostic bronchoalveolar lavage in critically ill mechanically ventilated patients. BMC Pulm Med. 2015 Sep 29;15:107. doi: 10.1186/s12890-015-0104-1. PMID 26420333
- [Background] Maitre B, Jaber S, Maggiore SM, Bergot E, Richard JC, Bakthiari H, Housset B, Boussignac G, Brochard L. Continuous positive airway pressure during fiberoptic bronchoscopy in hypoxemic patients. A randomized double-blind study using a new device. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):1063-7. doi: 10.1164/ajrccm.162.3.9910117. PMID 10988131
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Frat JP, Ragot S, Girault C, Perbet S, Prat G, Boulain T, Demoule A, Ricard JD, Coudroy R, Robert R, Mercat A, Brochard L, Thille AW; REVA network. Effect of non-invasive oxygenation strategies in immunocompromised patients with severe acute respiratory failure: a post-hoc analysis of a randomised trial. Lancet Respir Med. 2016 Aug;4(8):646-652. doi: 10.1016/S2213-2600(16)30093-5. Epub 2016 May 27. PMID 27245914
- [Background] Nishimura M. High-flow nasal cannula oxygen therapy in adults. J Intensive Care. 2015 Mar 31;3(1):15. doi: 10.1186/s40560-015-0084-5. eCollection 2015. PMID 25866645
- [Background] Lomas C, Roca O, Alvarez A, et al. Fibroscopy in patients with hypoxemic respiratory insufficiency: Utility of the high-flow nasal cannula. Respiratory Medicine CME 2009;2:121.
- [Background] Diab S, Fraser JF. Maintaining Oxygenation Successfully with High Flow Nasal Cannula during Diagnostic Bronchoscopy on a Postoperative Lung Transplant Patient in the Intensive Care. Case Rep Crit Care. 2014;2014:198262. doi: 10.1155/2014/198262. Epub 2014 Nov 13. PMID 25478241
- [Background] Miyagi K, Haranaga S, Higa F, Tateyama M, Fujita J. Implementation of bronchoalveolar lavage using a high-flow nasal cannula in five cases of acute respiratory failure. Respir Investig. 2014 Sep;52(5):310-4. doi: 10.1016/j.resinv.2014.06.006. Epub 2014 Jul 25. PMID 25169847
- [Background] 16. Kim KC, Hyun DS. Usefulness of high-flow nasal cannula (HFNC) oxygen delivery during bronchoalveolar lavage (BAL) in spontaneous breathing patients with hypoxemia. European Respiratory Journal. 2014; 44: p706.
- [Background] Lucangelo U, Vassallo FG, Marras E, Ferluga M, Beziza E, Comuzzi L, Berlot G, Zin WA. High-flow nasal interface improves oxygenation in patients undergoing bronchoscopy. Crit Care Res Pract. 2012;2012:506382. doi: 10.1155/2012/506382. Epub 2012 May 20. PMID 22666567
- [Background] Simon M, Braune S, Frings D, Wiontzek AK, Klose H, Kluge S. High-flow nasal cannula oxygen versus non-invasive ventilation in patients with acute hypoxaemic respiratory failure undergoing flexible bronchoscopy--a prospective randomised trial. Crit Care. 2014 Dec 22;18(6):712. doi: 10.1186/s13054-014-0712-9. PMID 25529351
- [Background] Parke R, McGuinness S, Eccleston M. Nasal high-flow therapy delivers low level positive airway pressure. Br J Anaesth. 2009 Dec;103(6):886-90. doi: 10.1093/bja/aep280. Epub 2009 Oct 20. PMID 19846404
- [Background] Antonelli M, Conti G, Rocco M, Arcangeli A, Cavaliere F, Proietti R, Meduri GU. Noninvasive positive-pressure ventilation vs. conventional oxygen supplementation in hypoxemic patients undergoing diagnostic bronchoscopy. Chest. 2002 Apr;121(4):1149-54. doi: 10.1378/chest.121.4.1149. PMID 11948045
- [Background] La Combe B, Messika J, Labbe V, Razazi K, Maitre B, Sztrymf B, Dreyfuss D, Fartoukh M, Ricard JD. High-flow nasal oxygen for bronchoalveolar lavage in acute respiratory failure patients. Eur Respir J. 2016 Apr;47(4):1283-6. doi: 10.1183/13993003.01883-2015. Epub 2016 Feb 11. No abstract available. PMID 26869676
- [Background] Fang WF, Chen YC, Chung YH, Woon WT, Tseng CC, Chang HW, Lin MC. Predictors of oxygen desaturation in patients undergoing diagnostic bronchoscopy. Chang Gung Med J. 2006 May-Jun;29(3):306-12. PMID 16924893
- [Background] 23. Chris Hau (respiratory therapist - Princess Margaret Hospital), Clodagh Ryan (Respirologist, Princess Margaret Hospital, Geeta Mehta (Respirologist, Princess Margaret Hospital) (personal communication, November 2016)
- [Background] Miguel-Montanes R, Hajage D, Messika J, Bertrand F, Gaudry S, Rafat C, Labbe V, Dufour N, Jean-Baptiste S, Bedet A, Dreyfuss D, Ricard JD. Use of high-flow nasal cannula oxygen therapy to prevent desaturation during tracheal intubation of intensive care patients with mild-to-moderate hypoxemia. Crit Care Med. 2015 Mar;43(3):574-83. doi: 10.1097/CCM.0000000000000743. PMID 25479117
- [Background] La Combe B, Messika J, Fartoukh M, Ricard JD. Increased use of high-flow nasal oxygen during bronchoscopy. Eur Respir J. 2016 Aug;48(2):590-2. doi: 10.1183/13993003.00565-2016. No abstract available. PMID 27478191
- [Background] Santos PS, Cruz C, Esquinas AM. Increased use of high-flow nasal oxygen during bronchoscopy. Eur Respir J. 2016 Aug;48(2):589. doi: 10.1183/13993003.00441-2016. No abstract available. PMID 27478190